CLINICAL TRIAL: NCT04330560
Title: Feasibility and Preliminary Evaluation and the Effects of Exercise-based Telerehabilitation on the Acceptability and Safety, and Clinical Effectiveness Among Patients With Coronary Heart Disease Undergoing the Cardiac Rehabilitation Program
Brief Title: Exercise-based Telerehabilitation in the Cardiac Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018112-6846; RF009C-2018 (Other Grant/Funding Number: University of Malaya Grant)
Record Dates: First submitted 2020-02-25; First posted 2020-04-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The masking will be imposed on the investigator who will be involved with the recruitment of the participant to prevent selection bias. The allocation of the participant to a group will be randomised using computer-generated random numbers by the other investigator who did not involve in recruiting the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ex group (Experimental): Receive CR telerehabilitation (exercise telemonitoring link to the healthcare platform + teleconsultation)
  Interventions: Device: Exercise telemonitoring connects to healthcare platform; Device: Exercise teleconsultation; Procedure: Other CR components
- Com group (Active Comparator): Receive CR telerehabilitation (exercise self-monitoring + teleconsultation)
  Interventions: Device: Exercise self-monitoring; Device: Exercise teleconsultation; Procedure: Other CR components
- C group (Placebo Comparator): Standard care - traditional center-based CR
  Interventions: Procedure: Standard care

INTERVENTIONS:
Device: Exercise telemonitoring connects to healthcare platform — The participant is required to wear the fitness tracker every day during waking hours throughout the 12 weeks of intervention (except during sleeping, bathing, and swimming) link to the healthcare practitioner
  Arms: Ex group
Device: Exercise self-monitoring — The participant is required to wear the fitness tracker every day during waking hours throughout the 12 weeks of intervention (except during sleeping, bathing, and swimming) for exercise self-monitoring.
  Arms: Com group
Device: Exercise teleconsultation — Conducted through smartphone video call app.
  Arms: Com group; Ex group
Procedure: Other CR components — Including dietary, psychology, education conducted at the center.
  Arms: Com group; Ex group
Procedure: Standard care — Undergoing standard care by cardiac rehabilitation at the center
  Arms: C group

SUMMARY:
The intervention will involve a system that comprises a wrist-worn activity tracker and a smartphone app that acts as a medium to link to the healthcare website

DETAILED DESCRIPTION:
Feasibility study objective: - To investigate the feasibility and preliminary of exercise-based telerehabilitation before undertaking full-scale RCT.

Randomized control trial objective: -

1. Primary Objective: To determine the exercise capacity among patients with CHD,
2. Secondary Objectives: To assess patient exercise adherence and determine the changes in other clinical health outcomes.

Study Population: Patients with coronary heart disease

Description of Sites/Facilities Enrolling Participants: Patient engagement with the cardiac rehabilitation phase 2 (CRP2) at the University Malaya Medical Centre (UMMC).

Description of Study Intervention: This study is a mixed-methods study consisting of a quantitative study (feasibility, preliminary evaluation, and full randomized control trial) and a qualitative study (interviewing). The present study will be conducting a single-blinded, three-arm, parallel over a 12-weeks study period during CRP2. Measurement will be collected during pre-and post-test.

ELIGIBILITY:
Inclusion Criteria:

* Adults with 18 years old and above with indexed diagnosis of coronary heart disease (CHD) and are referred for Cardiac Rehabilitation Program;
* Low- and moderate-risk patient category (controlled BP, sinus rhythm at 60-90 bpm, pain score< 3/10) and received a statement of medical clearance by a CR physician to undertake exercise with minimal supervision;
* The patient is willing to wear trackers during waking hours, own a personal smartphone and have access to internet/Wi-Fi; and
* Participant must be able to able to read, speak and understand English and Malay.

Exclusion Criteria:

* Heart failure NYHA Stage 3-4, pulse undetected by trackers;
* The participant who cannot detect their pulse through wrist-worn tracker;
* Do not own a smartphone with the mobile internet/Wi-Fi ; and
* Contraindicated for an exercise stress test and concomitant morbidity that limit physical activity and exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility (Recruitment procedure) | 12 weeks
  To inform the patient's acceptability towards recruitment procedure
Feasibility (Randomization procedure) | 12 weeks
  To inform the patient's acceptability towards randomization procedure
Feasibility (Cardiac rehabilitation program adherence) | 12 weeks
  To inform the patient's acceptability towards cardiac rehabilitation program adherence
Feasibility (Assessment adherence) | 12 weeks
  To inform the patient's acceptability towards assessment adherence
Feasibility (Safety - hospital readmission) | 12 weeks
  To inform the patient's safety on hospital readmission
Feasibility (Safety - cardiac adverse events) | 12 weeks
  To inform the patient's safety on cardiac adverse events
Exercise capacity during exercise stress test | 12 weeks
  Changes of metabolic equivalents (METs)
Exercise capacity during six-minutes walking test | 12 weeks
  Changes of walking distance (meter)

SECONDARY OUTCOMES:
Exercise adherence - Steps count | 12 weeks
  Changes in patient's weekly steps count.
Exercise adherence - Exercise frequency | 12 weeks
  Changes in patient's weekly exercise frequency.
Exercise adherence - Exercise duration | 12 weeks
  Changes in patient's weekly exercise duration (minutes).
Hospital readmission | 12 weeks
  Changes of frequency of hospital readmission throughout the intervention
Cardiac adverse events | 12 weeks
  Changes of frequency of cardiac adverse events throughout the intervention
Blood collection - serum cholesterol | 12 weeks
  Changes of serum cholesterol (mmol/L)
Blood collection - triglyceride | 12 weeks
  Changes of serum triglyceride (mmol/L)
Blood collection - high-density lipoproteins (HDL) | 12 weeks
  Changes of high-density lipoproteins (HDL) (mmol/L)
Blood collection - low-density lipoprotein (LDL) | 12 weeks
  Changes of low-density lipoprotein (LDL) (mmol/L)
Blood collection - Haemoglobin A1C (HA1c) | 12 weeks
  Changes of Haemoglobin A1C (HA1c) (mmols/mol)
Body mass (kg) | 12 weeks
  Changes of body mass (kg)
Body mass index (BMI) (kg/m2) | 12 weeks
  Changes of BMI (kg/m2)
Usability scale score | 12 weeks
  Measured by using mHealth App Usability Questionnaire (MAUQ). Indicators are evaluated according to the seven-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree" on smartphone app ease of use, interface and satisfaction, and usefulness.
Factors associated with non-adherence to cardiac rehabilitation program score | 12 weeks
  Measured by using Cardiac Rehabilitation Barriers Scale (CRBS) questionnaire. Indicators are evaluated according to the five-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree."
Quality of life (QOL) score | 12 weeks
  Measured by using WHO Quality of Life-BREF (WHOQOL-BREF) questionnaire. Indicators are evaluated according to the five-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree" on the physical health, psychological, social relationship and environment.
Fitness tracker acceptance score | 12 weeks
  Measured by using Technology Acceptance Model (TAM) questionnaire. Indicators are evaluated according to the five-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree" on the effort expectancy, performance expectancy, facilitating conditions, perceived enjoyment, perceived fee, perceived privacy, perceived trust, perceived value, social influence, perceived health increase and intention to use.
Participant's acceptance to the exercise-based telemonitoring | 12 weeks
  Exploring the participant's acceptance of the exercise-based telemonitoring through the interview session

CONTACTS AND LOCATIONS:
Overall Officials: Anwar Suhaimi, MBBS, Principal Investigator — University of Malaya; Wan Ling Lee, PhD, Principal Investigator — University of Malaya; Sanjay Rampal Lekhraj Rampal, PhD, Principal Investigator — University of Malaya
Locations (1):
- Rehabilitation Medicine, Pusat Perubatan Universiti Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536